CLINICAL TRIAL: NCT02455297
Title: A Single-arm, Open-label Phase IIa Study to Evaluate the Efficacy and Safety of Copanlisib Monotherapy in Patients With Relapsed or Refractory Mantle Cell Lymphoma (MCL), Who Failed Ibrutinib Treatment or Were Unable to Tolerate Ibrutinib
Brief Title: Phase IIa Study of Copanlisib in Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17120
Record Dates: First submitted 2015-05-23; First posted 2015-05-27 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Lymphoma, Mantle-Cell
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Copanlisib (Experimental): Copanlisib (BAY80-6946) solution for IV infusion
  Interventions: Drug: Copanlisib (BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (BAY80-6946) — Starting dose 60 mg (dose reduction due to toxicities to 45 mg allowed). Administered in slow IV bolus on days 1, 8 and 15 of each 28 day cycle until disease progression or until another criterion is met for withdrawal from study treatment.

SUMMARY:
The primary objective of this study is to assess objective response rate (ORR) in patients with relapsed or refractory MCL who failed ibrutinib treatment or were unable to tolerate ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed MCL
* Patients who have previously received treatment with ibrutinib (modified by amendment 1), including:

  * Completion of at least 1 cycle of treatment with ibrutinib and confirmed evidence of disease progression or refractoriness to treatment or
  * Discontinuation of ibrutinib treatment at an earlier time due to toxicity
* Measurable disease according to the Lugano Classification
* At least 28 days or 5 half-lives, whichever is shorter, from the completion of anti-cancer treatment (including, but not limited to, immunotherapy, chemotherapy, targeted therapy and biologic therapy) to the start of study treatment, excluding ibrutinib where the window may be less and at minimum 3 days (modified by amendment 1)
* Availability of fresh tumor tissue at screening
* Male or female patients ≥ 18 years old
* ECOG (Eastern Cooperative Oncology Group) performance status of ≤ 2
* Left ventricular ejection fraction (LVEF) by echocardiogram or multiple gated acquisition (MUGA) scan ≥ the lower limit of normal (LLN) for the Institution
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Any of the following as the only site(s) of disease: palpable lymph nodes not visible on imaging studies, skin lesions, or bone marrow involvement only
* Current central nervous system (CNS) involvement by lymphoma
* New York Heart Association (NYHA) class III or IV heart disease
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of study treatment
* Uncontrolled arterial hypertension despite optimal medical management (per investigator's assessment) (modified by amendment 1)
* Type I or II diabetes mellitus with HbA1c > 8.5% at screening (modified by amendment 1)
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before start of study treatment. However, if a patient has recovered to ECOG performance status of ≤ 2 he/she may be enrolled provided that other eligibility criteria are met
* Ongoing or active infection of Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 3
* Known history of human immunodeficiency virus (HIV) infection
* Acute or chronic hepatitis B (HBV) or hepatitis C (HCV) infection requiring concomitant treatment prohibited by this protocol (i.e.immunosuppressive therapy)
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
* Prior treatment with PI3K inhibitor(s)
* Cytomegalovirus (CMV) PCR positive at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 weeks
  ORR is defined as the proportion of patients who have a best overall response of complete response (CR) or partial response (PR) during study conduct according to the criteria defined by the Lugano response criteria in NHL 2014.

SECONDARY OUTCOMES:
Complete response rate (CRR) | 24 weeks
  Defined as the proportion of patients who have a best overall response of CR during study conduct according to the criteria defined by the Lugano response criteria in NHL 2014
Disease control rate (DCR) | 24 weeks
  Defined as the proportion of patients who have a best response of CR, PR, or stable disease (SD)
Progression-free survival (PFS) | 24 weeks
  Defined as the time (in days) from the date of first administration of study treatment to radiological disease progression or death from any cause (if death occurs before radiological progression is documented). PFS for patients without radiological progression or death at the time of analysis will be censored at the last date of evaluable tumor assessment. PFS for alive patients who have no tumor assessments after baseline will be censored at day 1.
Duration of response (DOR) | 24 weeks
  Defined as the time (in days) from the date of first observed tumor response of CR or PR, whichever was noted earlier, to radiological disease progression or death from any cause (if death occurs before radiological progression is documented)
Overall survival (OS) | 24 weeks
  Defined as the time (in days) from the date of first administration of study treatment to death from any cause. The OS time for patients alive at the time of analysis will be censored at their last known alive date.
Number of participants with treatment emergent adverse events (TEAEs) as a measure of safety and tolerability | Approximately 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- United States (4):
  - Baltimore, Maryland
  - Hackensack, New Jersey
  - New York, New York
  - Burlington, Vermont